CLINICAL TRIAL: NCT06457048
Title: Evaluation of a Locally Adapted Stroke Unit to Improve Outcomes in Lusaka, Zambia
Brief Title: Zambia Stroke Unit Study
Acronym: ZASUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00447874
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Outcomes will be compared between a prospective post-intervention cohort enrolled for this study and a historical pre-intervention cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke Unit Arm (Experimental): All participants in this study will be adults with stroke cared for in the recently implemented stroke unit at the University Teaching Hospital in Lusaka, Zambia. Of note, all adults with stroke admitted to the University Teaching Hospital during the study period will be cared for in the stroke unit regardless of participation participation in this study. However, only those who consent to study participation will have data collected.
  Interventions: Other: Stroke Unit
- Pre-Stroke Unit Arm (No Intervention): This arm will consist of a historical cohort of adults with stroke admitted to the University Teaching Hospital in Lusaka, Zambia for the implementation of a stroke unit.

INTERVENTIONS:
Other: Stroke Unit — The stroke unit at the University Teaching Hospital is a 12-bed unit on the general medical wards staffed by neurologists and nurses specifically trained in stroke care. This intervention includes new protocols and clinical practice guidelines that were developed by multiple stakeholders in Zambia to standardize stroke care, with a focus on early and consistent mobilization of patients with stroke, minimizing use of urinary catheters, provision of deep vein thrombosis prophylaxis, formal assessment of swallowing and assignment of modified diets as needed, and appropriate initiation of secondary prevention medications for stroke. Nurses and doctors working in this unit were trained on the new stroke unit protocols and are asked to follow these protocols in caring for patients with stroke admitted to the Stroke Unit.
  Arms: Stroke Unit Arm

SUMMARY:
The goal of this clinical trial is to evaluate the impact of a locally adapted stroke unit on outcomes of adults with stroke in Zambia. The main question[s] to answer are: • Does provision of evidence-based stroke care improve after implementation of a stroke unit at the University Teaching Hospital in Zambia? • Do patients cared for in a locally adapted stroke unit at the University Teaching Hospital in Zambia have better in-hospital and post-discharge outcomes that similar patients who were not cared for in the stroke unit? The investigators will collect data on the types of care participants receive during hospitalization and vital status (alive/dead) at the time of hospital discharge and at 90-days post-discharge. Researchers will compare patients enrolled in this study to a historical group of adults with stroke cared for at the same hospital prior to implementation of the stroke unit.

DETAILED DESCRIPTION:
The overarching goal of this project is to evaluate the uptake and impact of locally relevant, feasible, and generalizable stroke systems of care developed for the University Teaching Hospital (UTH) in Lusaka, Zambia using the Adopt-Contextualize-Adapt framework in order to improve stroke-related outcomes. Zambia is a country of ~20 million people in southern Africa where stroke is the eighth leading cause of death. However, stroke is not a problem unique to Zambia. Stroke is the second leading cause of adult disability and mortality worldwide. More than 75% of stroke-related morbidity and mortality occur in low- and middle-income countries (LMICs), and stroke prevalence in sub-Saharan Africa (SSA) is among the highest in the world. Yet, most stroke literature to date has been developed in high-income settings and its results applied to LMICs without adequate consideration of biological, ethnic, cultural and contextual differences. Diverse populations and settings in LMICs, including Zambia, necessitate evaluating unique risk factors, treatment strategies and systems of care in order to develop locally relevant interventions to improve stroke-related outcomes.

While acute stroke interventions (e.g., tissue plasminogen activator, endovascular therapies) have improved outcomes, indirect advances in stroke care have had a broader impact. Implementation of standardized systems of stroke care - i.e. stroke units - has led to secondary gains in stroke-related outcomes regardless of whether patients receive acute interventions. Compared to alternative care models, inpatient stroke unit care is associated with substantial reductions in death, dependency, and institutionalized care. In LMICs with limited access to specialists, neuroimaging, and acute stroke interventions, standardized systems of stroke care have not been instituted, including across Zambia and much of SSA. Absence of standardized systems of care likely accounts for higher rates of poor functional outcomes and mortality compared to higher-income settings.

Developing systems of stroke care in Zambia may improve stroke outcomes even in the absence of acute stroke interventions. Yet, simply instituting stroke clinical practice guidelines (CPGs) developed in high-income settings is unlikely to be successful without attention to differences in resource availability, health systems, and local contextual factors. Differences in biology (e.g. younger age, higher rates of HIV and rheumatic heart disease, differing risk factors) may also necessitate changes to stroke care delivery. As such, development of systems of stroke care in Zambia offers the promise of substantially improving stroke outcomes but must be done in a way in which stroke biology as well as cultural, patient, provider, and health systems factors are carefully considered during the design and implementation process.

Prior research characterized stroke care practices and stroke-related outcomes at the University Teaching Hospital (UTH) in Zambia. More recently, contextualized, locally relevant stroke CPGs were developed for UTH using the systematic guideline adaptation process of the Adopt-Contextualize-Adapt framework. These have recently been implemented as part of Zambia's first stroke unit. This project will assess the impact of local stroke CPGs on CPG adherence, stroke quality measures (QMs) and mortality through a post-intervention cohort of 300 adults with stroke. In this cohort, CPG uptake and in-hospital and post-discharge mortality will be measured and compared to a historical pre-intervention cohort of adults with stroke admitted to UTH before stroke unit implementation. If effective, results could potentially be applied across SSA thereby improving outcomes for millions of people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected diagnosis of stroke by treating neurologist or imaging-confirmed diagnosis of stroke
* Symptom onset (last known normal) within 7 days of presentation to the University Teaching Hospital in Lusaka, Zambia
* Inpatient admission to the University Teaching Hospital in Lusaka, Zambia

Exclusion Criteria:

* Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-08-17 (Actual)

PRIMARY OUTCOMES:
Proportion of clinical practice guidelines followed during inpatient admission | <=10 days of inpatient hospitalization for acute stroke (patients will be followed for the first 10 days of hospital admission or until hospital discharge, whichever is first)
  Whether or not each individual clinical practice guideline is followed will be tracked each day of the participant's inpatient admission for stroke. The total proportion of clinical practice guidelines followed will then be calculated.

SECONDARY OUTCOMES:
In-hospital mortality | Duration of inpatient hospitalization ( likely to average <7 days after enrollment ) up to 7 days
  Proportion of patients who die during the inpatient hospitalization for acute stroke
90-day post-discharge mortality | Duration of inpatient hospitalization + 90 days (likely to average < 100 days after enrollment)
  Proportion of patients who survive the inpatient hospitalization but die within 90 days of discharge as assessed by telephone call
Functional status at 90-days post-discharge | Duration of inpatient hospitalization + 90 days (likely to average <100 days after enrollment)
  Proportion of patients with Modified Rankin Scale (mRS) <2 vs mRS >=2 at 90-days post-discharge. mRS will be measured using the telephone version of the modified Rankin Scale and the study team will include all patients (not just those who survived the initial hospitalization) in this outcome.Score range from 0 to 6, with higher scores indicating greater disability.
Rate of aspiration pneumonia | <=10 days of inpatient hospitalization for acute stroke (patients will be followed for the first 10 days of hospital admission or until hospital discharge, whichever is first)
  Aspiration pneumonia will be defined as >=4 of the following criteria: fever (temperature >38°C), tachypnea (respiratory rate >20), hypoxemia (oxygen saturation <92%), cough, rhonchi, witnessed aspiration event, initiation of antibiotics for clinically suspected aspiration pneumonia, leukocytosis (WBC >10,000) on complete blood count (CBC) or opacity on chest X-ray. These criteria will be assessed daily for the first 10 days of admission or until discharge, whichever comes first.
Rate of decubitus ulcers | <=10 days of inpatient hospitalization for acute stroke (patients will be followed for the first 10 days of hospital admission or until hospital discharge, whichever is first)
  Presence or absence of decubitus ulcers will be assessed daily with a skin exam for the first ten days of inpatient hospitalization or until hospital discharge, whichever occurs first.
Rate of deep vein thrombosis | <=10 days of inpatient hospitalization for acute stroke (patients will be followed for the first 10 days of hospital admission or until hospital discharge, whichever is first)
  Proportion of patients diagnosed with a deep vein thrombosis confirmed on ultrasound during the first 10 days of hospitalization or until hospital discharge, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Saylor, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Study protocols and study materials as described below as well as a de-identified dataset will be shared if sharing criteria (described below) are met.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available one year after study completion for a period of three years.
Access Criteria: All requests for study data will need to be approved by the study team and by both a Zambian IRB (University of Zambia Biomedical Ethics Regulatory Committee or Excellence Research Ethics & Science (ERES) Converge IRB) and the Zambia National Health Research Authority prior to data sharing.